CLINICAL TRIAL: NCT00782535
Title: EVALUATION OF THE SAFETY AND EFFICACY OF TREATMENT WITH SINGLE DOSES OF CHF 4226 pMDI IN PATIENTS WITH CHRONIC OBSTRUCTIVE PULMONARY DISEASE A Multicenter, Randomized, Double-Blind,Placebo-Controlled, 5-Way Crossover Study
Brief Title: Safety and Efficacy Study of Treatment With Single Doses of CHF 4226 pMDI in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-0810-PR-0001
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A (Experimental): Single therapeutic dose of CHF 4226 pMDI
  Interventions: Drug: CHF 4226 pMDI
- Treatment B (Experimental): Single therapeutic dose of CHF 4226 pMDI
  Interventions: Drug: CHF 4226 pMDI
- Treatment C (Experimental): Single supratherapeutic dose of CHF 4226 pMDI
  Interventions: Drug: CHF 4226 pMDI
- Treatment D (Experimental): Single supratherapeutic dose of CHF 4226 pMDI
  Interventions: Drug: CHF 4226 pMDI
- Treatment E (Placebo Comparator): Single dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CHF 4226 pMDI — Inhaled solution, single therapeutic dose
  Arms: Treatment A; Treatment B
Drug: CHF 4226 pMDI — Inhaled solution, single supratherapeutic dose
  Arms: Treatment C; Treatment D
Drug: Placebo — Inhaled solution, single dose of placebo
  Arms: Treatment E

SUMMARY:
The purpose of this study is to characterize the dose-response profile of peak and trough FEV1 after single dose administrations of carmoterol in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed an IRB approved Informed Consent form and the written informed consent was obtained prior to any study-related procedure(s)
* Patient is a male or non-pregnant female, 40 -75 years old, inclusive
* Patient has a current or past cigarette smoking history of at least 15 pack-years
* Patient has a clinical diagnosis of COPD in accordance with the recommendations of the National Heart Lung and Blood Institute/World Health Organization (NHLBI/WHO) Global Initiative for Chronic Obstructive Lung Disease (GOLD)
* Patient meets the following requirements after an FEV1 albuterol reversibility test (i.e., 30 minutes following 400µg (metered dose) albuterol MDI):
* FEV1/FVC < 70%
* FEV1 is at least 0.9L
* FEV1 30% - 80%, inclusive, of patient's predicted normal value
* ∆FEV1 > 5% of pre-albuterol value
* If ∆FEV1 </= 5% of pre-albuterol value, then this requirement must be met after retesting during the run-in period, at least 24 hours prior to Visit 2.

Exclusion Criteria:

* Patient has a history of asthma
* Patient has a blood eosinophil count > 500/µL
* Patient has a history of allergic rhinitis or atopy
* Patient had a COPD exacerbation or a lower respiratory tract infection within 8 weeks prior to screening, or during the run-in period, that resulted in the use of an antibiotic, or oral or parenteral corticosteroids
* Patient is on an inhaled corticosteroid that has been initiated, or the effective dose has been changed, within 4 weeks prior to screening or during the run-in period
* Patient has an uncontrolled cardiovascular (e.g., uncontrolled hypertension), respiratory, hematologic, immunologic, renal, neurologic, hepatic, endocrine (e.g., uncontrolled diabetes mellitus) or other disease, or any condition that might, in the judgment of the Investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study
* Patient has clinically significant abnormal routine hematology (e.g., anemia) and/or clinical chemistry value(s).
* Patient has a history of coronary artery disease, cerebrovascular disease, cardiac arrhythmias
* Patient has lung cancer or a history of lung cancer
* Patient has active cancer or a history of cancer with less than 5 years disease free survival time (whether or not there is evidence of local recurrence or metastases). Localized basal cell carcinoma (without metastases) of the skin is acceptable.
* Patient has a serum potassium value ≤ 3.5 mEq/L or > 5.5mEq/L and/or a fasting serum glucose value ≥ 140 mg/dL
* Patient has an abnormal QTcF interval value in the Screening visit ECG test (i.e., > 450 msec in males or > 470 msec in females)
* Patient has developed Cor Pulmonale
* Patient is receiving long term oxygen therapy, i.e., > 16 hours/24-hour period, every day, unless residing at an elevation > 4000ft
* Patient has used any of the following medications prior to Screening and has not met the specified minimum washout period:
* Long acting anti-cholinergic agent (i.e., tiotropium): 7 days
* Short acting anti-cholinergics: 8 hours
* Fixed combinations of β2-agonists and inhaled corticosteroids: 48 hours
* Fixed combinations of an anti-cholinergic and short acting β2-agonist: 8 hours
* Long-acting β2-agonists: 48 hours
* Short acting β2-agonists: 6 hours
* Theophylline and other xanthines: 1 week
* Parenteral or oral corticosteroids: 1 month
* Patient has taken any non-permitted medication
* Patient has received a live-attenuated virus vaccination within two weeks prior to screening or during the run-in (inactivated Influenza vaccination is acceptable provided it is not administered within 48 hours prior to Screening)
* Patient has a known intolerance/hypersensitivity to β2-adrenergic agonists, propellant gases/excipients
* Patient is pregnant or lactating female, or female physiologically capable of becoming pregnant UNLESS they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL OR are using one or more of the following acceptable methods of contraception:
* surgical sterilization (e.g., bilateral tubal ligation, hysterectomy)
* hormonal contraception (implantable, patch, oral)
* double-barrier methods (any double combination of: IUD, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap)
* Patient is male and does not agree to use a medically acceptable contraceptive (abstain from sexual intercourse, or use a condom with spermicide), or has not had a vasectomy at least 6 months prior to study participation, unless their sexual partner is not of child-bearing potential
* Patient is mentally or legally incapacitated
* Patient has participated in another investigational study within 30 days prior to screening
* Patient abuses alcohol or other substances
* Patient does not maintain regular day/night, waking/sleeping cycles (e.g., night shift worker)
* Patient is potentially non-compliant or unable to perform required outcome measurements of the protocol

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
FEV1 | T-1hr, T-10min, and 15 and 30 minutes, 1, 2, 3, 23 and 24 hours for each treatment period

SECONDARY OUTCOMES:
serum potassium | pre dose and 1, 4, 6 and 24 hrs post dose for each treatment period
serum glucose | pre dose and 1, 4, 6 and 24 hrs post dose for each treatment period
plasma concentrations of CHF 4226 | pre dose and 15 minutes and 2 hours post dose for each treatment period
urinary excretion of CHF 4226 | pre dose and 0-24 hrs post dose for each treatment period
FVC | T-1hr, T-10min, and 15 and 30 minutes, 1, 2, 3, 23 and 24 hours for each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Gottschlich, MD, Principal Investigator — New Horizons Clinical Research
Locations (5):
- United States (5):
  - University Clinical Research DeLand, LLC, DeLand, Florida
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - New Horizons Clinical Research Center, Cincinnati, Ohio
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Spartanburg Medical Research, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: No